CLINICAL TRIAL: NCT02771743
Title: Response-based Treatment of High-risk Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-02-064
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Newly Diagnosed High Risk Neuroblastoma
Keywords: Neuroblastoma; High risk; Tandem high dose chemotherapy
MeSH Terms: conditions — Neuroblastoma | interventions — Cisplatin; Doxorubicin; Etoposide; Cyclophosphamide; Ifosfamide; Carboplatin; Radiotherapy; Interleukin-2; Isotretinoin; 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High risk neuroblastoma (Experimental): 1. Nine cycles of induction chemotherapy with cisplatin, etoposide, doxorubicin, cyclophosphamide (CEDC) and ifosfamide, carboplatin, etoposide (ICE) regimen
  2. Upfront surgery or surgery after 6 cycles of chemotherapy
  3. Peripheral stem cell mobilization after 7 cycles of chemotherapy
  4. Tandem high dose chemotherapy with autologous stem cell transplantation (Tandem HDCT/auto-SCT)
     * Dose of chemotherapeutic agents of 1st HDCT is tailored according to the residual positron emission tomography (PET)/Metaiodobenzylguanidine (MIBG) uptake before 1st HDCT
     * Dose of MIBG of 2nd HDCT is tailored according to the residual PET/MIBG uptake before 2nd HDCT
  5. Radiotherapy after tandem HDCT
  6. Immunotherapy and differentiation therapy with Interleukin-2/isotretinoin
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Ifosfamide; Drug: Carboplatin; Procedure: Tandem HDCT/auto-SCT; Radiation: Radiotherapy; Drug: Interleukin-2; Drug: Isotretinoin; Radiation: MIBG

INTERVENTIONS:
Drug: Cisplatin
Drug: Doxorubicin
Drug: Etoposide
Drug: Cyclophosphamide
Drug: Ifosfamide
Drug: Carboplatin
Procedure: Tandem HDCT/auto-SCT
Radiation: Radiotherapy
Drug: Interleukin-2
Drug: Isotretinoin
Radiation: MIBG

SUMMARY:
The purpose of this study is to improve outcome of high risk neuroblastoma by tailoring the treatment intensity of tandem high dose chemotherapy according to the treatment response to induction chemotherapy.

DETAILED DESCRIPTION:
Although the outcome of high-risk neuroblastoma improved after the introduction of high-dose chemotherapy and autologous stem cell transplantation (HDCT/autoSCT), the outcome still needs to be unsatisfactory.

In the investigator's previous study, good responders who had greater reduction of tumor volume after induction chemotherapy showed lower relapse-free survival compared to poor responders.Simultaneously, the reduction in tumor volume also was greater in patients who died of treatment related mortality than patients who had relapsed tumors. These findings suggest that tailoring treatment intensity according to the early tumor response to induction chemotherapy may improve patient outcomes. So, in this study investigators tailored the treatment intensity of high dose chemotherapy according to the treatment response to induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed high risk neuroblastoma
* Patients with informed consent

Exclusion Criteria:

* Patients with progressive disease or relapse
* Patients who underwent high dose chemotherapy before
* Patients with organ dysfunction as follows (creatinine elevation > 3 x upper limit of normal, Total bilirubin > 3 x upper limit of normal, aspartate transaminase/alanine transaminase > 5 x upper limit of normal), ejection fraction <40%
* Pregnant or nursing women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Rate of event free survival | Up to 3 years

SECONDARY OUTCOMES:
Rate of late adverse effects | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Sung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea